CLINICAL TRIAL: NCT01837589
Title: Evaluation of the Bone Mineralization by Quantitative Computed Tomodensitometry in Patients With Cystic Fibrosis : Validation Study
Brief Title: Quantitative Computed Tomodensitometry in Patients With Cystic Fibrosis
Acronym: TOMODENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Necker-Enfants Malades (Other)
Collaborators: Vaincre la Mucoviscidose (Other)
Responsible Party: Principal Investigator, Isabelle Sermet-Gaudelus, Professor, Hôpital Necker-Enfants Malades
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: N° ID RCB : 2009-A00292-55
Record Dates: First submitted 2012-11-15; First posted 2013-04-23 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis-DXA-QCT-Osteopenia- Osteoporosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- QCT and DXA (Other): All the patients will have both QCT and DXA
  Interventions: Other: QCT; Other: DXA

INTERVENTIONS:
Other: QCT
  Other Names: Quantitative Computed Tomodensitometry
Other: DXA
  Other Names: Dual-emission X-ray

SUMMARY:
The purpose of this study is to conduct a comparative study for the study of bone mineralization evaluated with Quantitative computed tomodensitometry (QCT) compared to the reference technique, Dual-emission X-ray absorptiometry (DXA).

DETAILED DESCRIPTION:
Patients with cystic fibrosis can have a deficit in bone mineralization. This is particularly well described in adults. However, in the pediatric population the results are more heterogeneous. The evaluation is hindered by difficulties in standardization of DXA interpretation.

This measurement depends from the mass and size of the bone as well as the mass of soft tissue covering the bone area. These two characteristics, intrinsic to the measurement, pose a significant problem of interpretations in children because a change in bone density may reflect both a change in bone mineral content or changes related to growth, for example, the increase in bone size or volume of soft tissue covering the bone of interest.

Quantitative computed tomography (QCT) provides a direct measure of bone mineralization densitometry volume. It quantifies bone mineral content in relation to the volume of the bone, in reference to an external phantom. This method therefore overcomes the size size.

This technique can be considered without an additional radiation exposure to patients during a lung CT because it is usual that lumbar vertebrae are included in the measurement window because of pulmonary hyperinflation. This exam would be ideal for patients with Cystic fibrosis.

All patients have these two evaluations during their routine management. This study compare study on the bone mineralization evaluated by (QCT) compared to the reference technique by (DXA) for the patient affected by cystic fibrosis for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by cystic fibrosis
* Aged over 5 years
* Patients whose clinical condition warrants an indication of chest CT in relation to the criteria of the french consensus conference on Cystic fibrosis in May 2002 (Palace of the Luxembourg).
* Patients whose clinical condition warrants an indication of DXA examination in accordance with French recommendations (Consensus of the Working Group "bone mineralization and cystic fibrosis" In children, the examination is recommended for ages 8 every 2 years if the Z-score is greater than - 1, every year if the Z-score is less than - 1.. In adults, the exam is recommended every 5 years if the T-score is greater than> - 1, every 2 years if it is between -1 and - 2; annually if less than - 2.)
* Patient does not exhibit a phase of bronchial exacerbation
* Collection of non-opposition of the patient
* Patient affiliated to social security

Exclusion Criteria:

* Patient transplanted
* Patient with an infective exacerbation phase

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of the mineralization with DXA(Dual-energy X-ray absorptiometry) as a Zscore of Bone mineral density and the Zscore of QCT (Quantitative computed tomography) | 1 day
  Evaluation of the mineralization with DXA(Dual-energy X-ray absorptiometry) as a Zscore of Bone mineral density(reference population: same sex, same bone age) and the Zscore of QCT (Quantitative computed tomography) (reference population: same sex, same age)

SECONDARY OUTCOMES:
Evaluation of the prevalence of osteopenia in children and adult affected by cystic fibrosis. | 1 day
Correlation of bone mineralization with nutritional status (BMI) | 1 day
Correlation of bone mineralization with respiratory status (FEV % predicted) | 1 day
Correlation of bone mineralization with Vitamine D (25(OH)vitD) | 1 day
Correlation of bone mineralization with the amount of total inhaled and oral corticosteroids administered (total number of days of steroids according to diiferent modalities: inhaled, oral IV) | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Sermet-Gaudelus, Professor, Principal Investigator — Necker Hospital
Locations (1):
- Necker Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No